CLINICAL TRIAL: NCT03619538
Title: Interest of the Nefopam and PCA Morphine Combination for Postoperative Analgesia in Patients Undergoing Colon Surgery
Acronym: NEFOPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-I/2003/JYL-01
Record Dates: First submitted 2018-07-25; First posted 2018-08-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2018-08

CONDITIONS: Colonic Neoplasms; Diverticulosis, Colonic
MeSH Terms: conditions — Colonic Neoplasms; Diverticulosis, Colonic | interventions — Nefopam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Other: saline solution
- Nefopam group (Experimental)
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam — The nefopam group received 120 mg nefopam (Acupan, Pharmbio, France) by continuous iv infusion over the study period (48h)
  Arms: Nefopam group
Other: saline solution — The Control group received 120 mg placebo infusion (saline solution) by continuous iv infusion over the study period (48h).
  Arms: control group

SUMMARY:
This study analyses interest of iv nefopam in combination with paracetamol after major abdominal surgery because the effect of morphine-sparing is discussed when combined these agents.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with a score ASA between I and III
* Patient scheduled for elective major abdominal surgery (by laparotomy) for cancer or diverticulosis
* Patient that signed the consent form

Exclusion Criteria:

* - Patient treated in emergency situation
* Patient with chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Patient that needs a surgery for restoration of continuity
* Patient pregnant, breastfeeding, or during periods of genital activity using no contraception.
* Patient with contraindications to nefopam, morphine, or paracetamol
* Patient with chronic obstructive pulmonary disease, renal or severe hepatic impairment
* Patient under analgesics treatment
* Patient who participated in a clinical study in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2007-06-25 (Actual); Study Completion 2007-06-25 (Actual)

PRIMARY OUTCOMES:
Estimate morphine consumption | over 48 hours
  mg

CONTACTS AND LOCATIONS:
Overall Officials: Jacques RIPART, Dr, Principal Investigator — Nîmes University Hospital

REFERENCES:
- [Result] Cuvillon P, Zoric L, Demattei C, Alonso S, Casano F, L'hermite J, Ripart J, Lefrant JY, Muller L. Opioid-sparing effect of nefopam in combination with paracetamol after major abdominal surgery: a randomized double-blind study. Minerva Anestesiol. 2017 Sep;83(9):914-920. doi: 10.23736/S0375-9393.17.11508-7. Epub 2017 Feb 13. PMID 28192892